CLINICAL TRIAL: NCT00767286
Title: A PHASE III TRIAL OF THE USE OF LONG TERM TOTAL ANDROGEN SUPPRESSION FOLLOWING NEOADJUVANT HORMONAL CYTOREDUCTION AND RADIOTHERAPY IN LOCALLY ADVANCED CARCINOMA OF THE PROSTATE
Brief Title: Goserelin, Flutamine, and Radiation Therapy in Treating Patients With Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077690; RTOG-9202
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2011-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin

INTERVENTIONS:
Drug: flutamide
Drug: goserelin acetate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Patient abstract not available

PURPOSE: Patient abstract not available

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare locoregional control, disease-free survival, and overall survival in patients with carcinoma of the prostate who are considered at high risk of relapse and receive long-term adjuvant zoladex (ZDX) vs. no adjuvant treatment following neoadjuvant ZDX/flutamide and radiotherapy. II. Compare sexual function in patients treated with these two regimens.

OUTLINE: Randomized study. Arm I: Neoadjuvant Antiandrogen Therapy and Releasing Factor Agonist Therapy plus Radiotherapy. Flutamide, FLUT, NSC-147834; and Zoladex, ZDX, NSC-606864; plus external-beam irradiation using megavoltage equipment with energies of at least 4 MV (at least 6 MV preferred). Arm II: Neoadjuvant Antiandrogen Therapy and Releasing Factor Agonist Therapy plus Radiotherapy followed by Adjuvant Releasing Factor Agonist Therapy. FLUT; and ZDX; plus external-beam irradiation using equipment as in Arm I; followed by ZDX.

PROJECTED ACCRUAL: 1,508 patients will be accrued over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, locally advanced adenocarcinoma of the prostate, including: Bulky primary tumors confined to the prostate (clinical Stage T2c) Primary tumors extending beyond the capsule (clinical Stage T3-4) No common iliac or para-aortic nodal involvement Regional lymph node involvement below the common iliac level allowed Positive nodes on imaging studies must be biopsied by FNA or surgical sampling PSA no more than 150 (mandatory) No distant metastases

PATIENT CHARACTERISTICS: Age: At least 50 Performance status: Karnofsky 70-100% Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No prior or concurrent second cancer except basal cell skin cancer No major medical or psychiatric illness that would prevent completion of treatment or interfere with follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No prior hormonal therapy Radiotherapy: No prior radiotherapy Surgery: No prior radical surgery for carcinoma of the prostate

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald E. Hanks, MD, Study Chair — Fox Chase Cancer Center

REFERENCES:
- [Background] Du KL, Bae K, Movsas B, Yan Y, Bryan C, Bruner DW. Impact of marital status and race on outcomes of patients enrolled in Radiation Therapy Oncology Group prostate cancer trials. Support Care Cancer. 2012 Jun;20(6):1317-25. doi: 10.1007/s00520-011-1219-4. Epub 2011 Jul 1. PMID 21720747
- [Background] Hamstra DA, Bae K, Pilepich MV, Hanks GE, Grignon DJ, McGowan DG, Roach M, Lawton C, Lee RJ, Sandler H. Older age predicts decreased metastasis and prostate cancer-specific death for men treated with radiation therapy: meta-analysis of radiation therapy oncology group trials. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1293-301. doi: 10.1016/j.ijrobp.2010.07.2004. Epub 2011 Mar 31. PMID 21458924
- [Background] Rodrigues G, Bae K, Roach M, Lawton C, Donnelly B, Grignon D, Hanks G, Porter A, Lepor H, Sandler H. Impact of ultrahigh baseline PSA levels on biochemical and clinical outcomes in two Radiation Therapy Oncology Group prostate clinical trials. Int J Radiat Oncol Biol Phys. 2011 Jun 1;80(2):445-52. doi: 10.1016/j.ijrobp.2010.02.034. Epub 2010 Aug 24. PMID 20615632
- [Background] Roach M 3rd, Bae K, Lawton C, Donnelly BJ, Grignon D, Hanks GE, Porter A, Lepor H, Venketesan V, Sandler H. Baseline serum testosterone in men treated with androgen deprivation therapy and radiotherapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Dec 1;78(5):1314-22. doi: 10.1016/j.ijrobp.2009.09.073. Epub 2010 Apr 8. PMID 20378270
- [Background] Roach M 3rd, Waldman F, Pollack A. Predictive models in external beam radiotherapy for clinically localized prostate cancer. Cancer. 2009 Jul 1;115(13 Suppl):3112-20. doi: 10.1002/cncr.24348. PMID 19544539
- [Background] Lawton CA, Bae K, Pilepich M, Hanks G, Shipley W. Long-term treatment sequelae after external beam irradiation with or without hormonal manipulation for adenocarcinoma of the prostate: analysis of radiation therapy oncology group studies 85-31, 86-10, and 92-02. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):437-41. doi: 10.1016/j.ijrobp.2007.06.050. Epub 2007 Sep 19. PMID 17881145
- [Background] Lawton CA, Michalski J, El- Naqa I, et al.: RTOG: genitourinary radiation oncology specialists reach consensus on pelvic lymph node volumes for high risk prostate cancer. [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-6, 2008.
- [Background] Whelan P. Editorial comment on: Cardiovascular mortality and duration of androgen deprivation for locally advanced prostate cancer: analysis of RTOG 92-02. Eur Urol. 2008 Oct;54(4):823-4. doi: 10.1016/j.eururo.2008.01.022. Epub 2008 Jan 15. No abstract available. PMID 18243509
- [Background] Paner GP, Bae K, Grignon DJ, et al.: Trends in Gleason grading of prostate cancer (PCa): analysis of reporting by institutional and central review pathologists in four Radiation Therapy Oncology Group (RTOG) protocols spanning 17 years and 2094 needle biopsies (bxs). [Abstract] United States and Canadian Academy of Pathology 96th Annual Meeting, March 24-30, 2007, San Diego, CA. A-766, 2007.
- [Background] Hachem P, Bae K, Khor L, et al.: Prostate tumor biomarker stability in archival tissue from men treated with radiotherapy: an analysis of RTOG 92-02 and Fox Chase randomized trials. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2280, S365-6, 2006.
- [Background] Lawton CA, Bae K, Pilepich M, et al.: Long-term treatment sequelae following external beam irradiation + hormonal manipulation for adenocarcinoma of the prostate: analysis of RTOG studies 85-31, 86-10, and 92-02. [Abstract] 2006 Prostate Cancer Symposium, February 24-26, 2006, San Francisco, CA. A-191, 2006.
- [Background] Pan CC, Bae K, Hanks GE, et al.: Comparison of two types of biochemical failures within the ASTRO and Phoenix Consensus definitions in patients treated on RTOG 92-02 and 94-13. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2196, S318, 2006.
- [Background] Pollack A, Bae K, Khor LY, et al.: Stability of tumor biomarkers in archival tissue from men treated with radiotherapy for prostate cancer: an analysis of RTOG 92-02 and Fox Chase randomized trials. [Abstract] Int J Biol Markers 22 (1): 72-3, 2006.
- [Background] Roach M, Moughan J, Movsas B, et al.: Socio-demographic predictors of biochemical failure and survival among high risk patients treated on Radiation Therapy Oncology Group (RTOG) prostate cancer trials: a meta-analysis. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1127, S204, 2006.
- [Result] Khor LY, Bae K, Paulus R, Al-Saleem T, Hammond ME, Grignon DJ, Che M, Venkatesan V, Byhardt RW, Rotman M, Hanks GE, Sandler HM, Pollack A. MDM2 and Ki-67 predict for distant metastasis and mortality in men treated with radiotherapy and androgen deprivation for prostate cancer: RTOG 92-02. J Clin Oncol. 2009 Jul 1;27(19):3177-84. doi: 10.1200/JCO.2008.19.8267. Epub 2009 May 26. PMID 19470936
- [Result] Pollack A, Bae K, Khor LY, Al-Saleem T, Hammond ME, Venkatesan V, Byhardt RW, Asbell SO, Shipley WU, Sandler HM. The importance of protein kinase A in prostate cancer: relationship to patient outcome in Radiation Therapy Oncology Group trial 92-02. Clin Cancer Res. 2009 Sep 1;15(17):5478-84. doi: 10.1158/1078-0432.CCR-08-2704. Epub 2009 Aug 25. PMID 19706804
- [Result] Ray ME, Bae K, Hussain MH, Hanks GE, Shipley WU, Sandler HM. Potential surrogate endpoints for prostate cancer survival: analysis of a phase III randomized trial. J Natl Cancer Inst. 2009 Feb 18;101(4):228-36. doi: 10.1093/jnci/djn489. Epub 2009 Feb 10. PMID 19211454
- [Result] Efstathiou JA, Bae K, Shipley WU, Hanks GE, Pilepich MV, Sandler HM, Smith MR. Cardiovascular mortality and duration of androgen deprivation for locally advanced prostate cancer: analysis of RTOG 92-02. Eur Urol. 2008 Oct;54(4):816-23. doi: 10.1016/j.eururo.2008.01.021. Epub 2008 Jan 15. PMID 18243498
- [Result] Horwitz EM, Bae K, Hanks GE, Porter A, Grignon DJ, Brereton HD, Venkatesan V, Lawton CA, Rosenthal SA, Sandler HM, Shipley WU. Ten-year follow-up of radiation therapy oncology group protocol 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol. 2008 May 20;26(15):2497-504. doi: 10.1200/JCO.2007.14.9021. Epub 2008 Apr 14. PMID 18413638
- [Result] Smith MR, Bae K, Efstathiou JA, Hanks GE, Pilepich MV, Sandler HM, Shipley WU. Diabetes and mortality in men with locally advanced prostate cancer: RTOG 92-02. J Clin Oncol. 2008 Sep 10;26(26):4333-9. doi: 10.1200/JCO.2008.16.5845. PMID 18779620
- [Result] Chakravarti A, DeSilvio M, Zhang M, Grignon D, Rosenthal S, Asbell SO, Hanks G, Sandler HM, Khor LY, Pollack A, Shipley W; Radiation Therapy Oncology Group. Prognostic value of p16 in locally advanced prostate cancer: a study based on Radiation Therapy Oncology Group Protocol 9202. J Clin Oncol. 2007 Jul 20;25(21):3082-9. doi: 10.1200/JCO.2006.08.4152. PMID 17634487
- [Result] Khor LY, Bae K, Pollack A, Hammond ME, Grignon DJ, Venkatesan VM, Rosenthal SA, Ritter MA, Sandler HM, Hanks GE, Shipley WU, Dicker AP. COX-2 expression predicts prostate-cancer outcome: analysis of data from the RTOG 92-02 trial. Lancet Oncol. 2007 Oct;8(10):912-20. doi: 10.1016/S1470-2045(07)70280-2. Epub 2007 Sep 18. PMID 17881290
- [Result] Khor LY, Moughan J, Al-Saleem T, Hammond EH, Venkatesan V, Rosenthal SA, Ritter MA, Sandler HM, Hanks GE, Shipley WU, Pollack A. Bcl-2 and Bax expression predict prostate cancer outcome in men treated with androgen deprivation and radiotherapy on radiation therapy oncology group protocol 92-02. Clin Cancer Res. 2007 Jun 15;13(12):3585-90. doi: 10.1158/1078-0432.CCR-06-2972. PMID 17575222
- [Result] Ray ME, Bae K, Hussain MHA, et al.: Surrogate endpoints for prostate cancer survival: a secondary analysis of RTOG 9202. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-143, S81-82, 2007.
- [Result] Roach M 3rd, De Silvio M, Rebbick T, Grignon D, Rotman M, Wolkov H, Fisher B, Hanks G, Shipley WU, Pollack A, Sandler H, Watkins-Bruner D. Racial differences in CYP3A4 genotype and survival among men treated on Radiation Therapy Oncology Group (RTOG) 9202: a phase III randomized trial. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):79-87. doi: 10.1016/j.ijrobp.2007.03.008. Epub 2007 May 10. PMID 17498886
- [Result] Hanks GE, Bae K, Porter AT, et al.: Ten year follow-up of RTOG 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-22, S13, 2006.
- [Result] Khor L, Bae K, Hammond ME, et al.: Cox-2 overexpression predicts prostate cancer outcome: an analysis of RTOG 92-02. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1124, S202, 2006.
- [Result] Khor LY, Bae K, Hammond ME, et al.: COX-2 overexpression in pretreatment diagnostic tissue is associated with prostate cancer outcome in RTOG 92-02. [Abstract] Int J Biol Markers 22 (1): 73-4, 2006.
- [Result] Konski A, Watkins-Bruner D, Brereton H, Feigenberg S, Hanks G. Long-term hormone therapy and radiation is cost-effective for patients with locally advanced prostate carcinoma. Cancer. 2006 Jan 1;106(1):51-7. doi: 10.1002/cncr.21575. PMID 16323171
- [Result] Valicenti RK, DeSilvio M, Hanks GE, Porter A, Brereton H, Rosenthal SA, Shipley WU, Sandler HM; Radiation Therapy Oncology Group Protocol 92-02. Posttreatment prostatic-specific antigen doubling time as a surrogate endpoint for prostate cancer-specific survival: an analysis of Radiation Therapy Oncology Group Protocol 92-02. Int J Radiat Oncol Biol Phys. 2006 Nov 15;66(4):1064-71. doi: 10.1016/j.ijrobp.2006.06.017. Epub 2006 Sep 18. PMID 16979837
- [Result] Khor LY, Desilvio M, Li R, McDonnell TJ, Hammond ME, Sause WT, Pilepich MV, Okunieff P, Sandler HM, Pollack A. Bcl-2 and bax expression and prostate cancer outcome in men treated with radiotherapy in Radiation Therapy Oncology Group protocol 86-10. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):25-30. doi: 10.1016/j.ijrobp.2006.03.056. Epub 2006 Jul 11. PMID 16814949
- [Result] Pollack A, Moughan J, Khor LY, et al.: BCL-2 and BAX are determinants of prostate cancer outcome in men treated with androgen deprivation and radiotherapy on RTOG 92-02. [Abstract] Int J Biol Markers 22 (1): 79, 2006.
- [Result] Chakravarti A, DeSilvio M, Zhang M, et al.: The prognostic value of p16 expression in locally advanced prostate cancer: a study based on RTOG 92-02. [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-30, S17, 2005.
- [Result] Che M, DeSilvio M, Pollack A, Grignon DJ, Venkatesan VM, Hanks GE, Sandler HM; RTOG. Prognostic value of abnormal p53 expression in locally advanced prostate cancer treated with androgen deprivation and radiotherapy: a study based on RTOG 9202. Int J Radiat Oncol Biol Phys. 2007 Nov 15;69(4):1117-23. doi: 10.1016/j.ijrobp.2007.04.070. Epub 2007 Aug 8. PMID 17689883
- [Result] Pollack A, DeSilvio M, Khor L, et al.: MDM2 expression is independent of P53 and Ki-67 in predicting prostate cancer outcome: an analysis of RTOG 92-02. [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-29, S17, 2005.
- [Result] Pollack A, DeSilvio M, Khor LY, Li R, Al-Saleem TI, Hammond ME, Venkatesan V, Lawton CA, Roach M 3rd, Shipley WU, Hanks GE, Sandler HM. Ki-67 staining is a strong predictor of distant metastasis and mortality for men with prostate cancer treated with radiotherapy plus androgen deprivation: Radiation Therapy Oncology Group Trial 92-02. J Clin Oncol. 2004 Jun 1;22(11):2133-40. doi: 10.1200/JCO.2004.09.150. PMID 15169799
- [Result] Hanks GE, Pajak TF, Porter A, Grignon D, Brereton H, Venkatesan V, Horwitz EM, Lawton C, Rosenthal SA, Sandler HM, Shipley WU; Radiation Therapy Oncology Group. Phase III trial of long-term adjuvant androgen deprivation after neoadjuvant hormonal cytoreduction and radiotherapy in locally advanced carcinoma of the prostate: the Radiation Therapy Oncology Group Protocol 92-02. J Clin Oncol. 2003 Nov 1;21(21):3972-8. doi: 10.1200/JCO.2003.11.023. PMID 14581419
- [Result] Pollack A, DeSilvio M, Khor L, et al.: Ki-67 staining is a strong predictor of patient outcome for prostate cancer patients treated with androgen deprivation plus radiotherapy: an analysis of RTOG 92-02. [Abstract] Int J Radiat Oncol Biol Phys 57 (2 Suppl): S200-1, 2003.
- [Result] Sandler HM, Pajak TF, Hanks GE, et al.: Can biochemical failure (ASTRO definition) be used as a surrogate endpoint for prostate cancer survival in phase III localized prostate cancer clinical trials? Analysis of RTOG protocol 92-02. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1529, 2003.
- [Result] Hanks GE, Lu JD, Machtay M, et al.: RTOG protocol 92-02: a phase III trial of the use of long term total androgen supppression following neoadjuvant hormonal cytoreduction and radiotherapy in locally advanced carcinoma of the prostate. [Abstract] Int J Radiat Oncol Biol Phys 48 (3 suppl): A-4, 112, 2000.
- [Derived] Armstrong AJ, Liu VYT, Selvaraju RR, Chen E, Simko JP, DeVries S, Sartor O, Sandler HM, Mohamad O, Huang HC, Griffin J, Yamashita R, Esteva A, Tran PT, Spratt DE, Carson JH, Peters C, Gore E, Lee SP, Monson JM, Augspurger ME, El-Gayed A, Rodgers JP, McKay R, Morgan T, Feng FY, Nguyen PL. Development and Validation of an Artificial Intelligence Digital Pathology Biomarker to Predict Benefit of Long-Term Hormonal Therapy and Radiotherapy in Men With High-Risk Prostate Cancer Across Multiple Phase III Trials. J Clin Oncol. 2025 Nov 10;43(32):3494-3504. doi: 10.1200/JCO.24.00365. Epub 2025 Apr 16. PMID 40239134
- [Derived] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143
- [Derived] Nguyen PL, Huang HR, Spratt DE, Davicioni E, Sandler HM, Shipley WU, Efstathiou JA, Simko JP, Pollack A, Dicker AP, Roach M, Rosenthal SA, Zeitzer KL, Mendez LC, Hartford AC, Hall WA, Desai AB, Rabinovitch RA, Peters CA, Rodgers JP, Tran P, Feng FY. Analysis of a Biopsy-Based Genomic Classifier in High-Risk Prostate Cancer: Meta-Analysis of the NRG Oncology/Radiation Therapy Oncology Group 9202, 9413, and 9902 Phase 3 Randomized Trials. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):521-529. doi: 10.1016/j.ijrobp.2022.12.035. Epub 2022 Dec 31. PMID 36596347